CLINICAL TRIAL: NCT00662519
Title: Short Course of Pegylated GCSF (Neulasta®) as Immunomodulatory Therapy for Type 1 Diabetes
Brief Title: Neulasta in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UF IRB 280-2006; JDRF 11-2007-825 (Other Grant/Funding Number: JDRF); 1R21DK078863-01A1 (NIH); GCRC 683 (Other Grant/Funding Number: GCRC)
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pegfilgrastim; pegylated granulocyte colony-stimulating factor; Sodium Chloride; Hematologic Tests; Hemoglobin A; Human Papillomavirus DNA Tests; HLA Antigens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neulasta (Experimental): Subjects will receive Neulasta subcutaneously every 2 weeks for 12 weeks (6 doses). In addition, the following test will be done: Mixed Meal Tolerance Test (MMTT), Hemoglobin A1C (HbA1c) blood test, and Human Leukocyte Antigen (HLA) DNA Test.
  Interventions: Drug: Neulasta (Pegylated); Dietary Supplement: Mixed Meal Tolerance Test (MMTT); Other: Blood test; Other: DNA Test
- Placebo (Placebo Comparator): Placebo injections will be given in identical volumes in identical syringes in the identical subcutaneous manner. In addition, the following test will be done: Mixed Meal Tolerance Test (MMTT), Hemoglobin A1C (HbA1c) blood test, and Human Leukocyte Antigen (HLA) DNA Test.
  Interventions: Drug: Placebo; Dietary Supplement: Mixed Meal Tolerance Test (MMTT); Other: Blood test; Other: DNA Test

INTERVENTIONS:
Drug: Neulasta (Pegylated) — Subjects will receive 6mg/dose given every 2 weeks for 12 weeks. Subjects less than 45kg will receive 100mcg/kg/dose every 2 weeks for 12 weeks.
  Other Names: Pegylated granulocyte colony stimulating factor (GCSF)
  Arms: Neulasta
Drug: Placebo — Placebo injections will be given in identical volumes in identical syringes in the identical subcutaneous manner. 6mg/dose given every 2 weeks for 12 weeks. Subjects less than 45kg will receive 100mcg/kg/dose every 2 weeks for 12 weeks.
  Other Names: Saline
  Arms: Placebo
Dietary Supplement: Mixed Meal Tolerance Test (MMTT) — This is a 2 hour test to find out how much C-peptide is being produced. C-peptide is used to measure the insulin being made by the cells of the pancreas. Both groups will have this test performed.
Other: Blood test — HbA1c is a blood test that measures the average blood sugar control and will be performed in both groups.
  Other Names: Hemoglobin A1C (HbA1c)
Other: DNA Test — The HLA test looks at the different chromosomes (DNA) for diabetes and will be performed in both groups.
  Other Names: Human Leukocyte Antigen (HLA)

SUMMARY:
The primary purpose of this study is to find out if giving a 12 week course of Neulasta (Pegylated granulocyte colony stimulating factor (GCSF)) to people with type 1 diabetes (T1D) is safe. The secondary purpose of this research study is to determin if giving GCSF to patients with T1D changes the immune system or preserves insulin production.

DETAILED DESCRIPTION:
As a participant in this study the following will happen:

Blood test, Mixed meal Tolerance Test (MMT) to find out how much C-peptide is being produced, Human Leukocyte Antigen (HLA) test, Hemoglobin A1C (HbA1c) test for overall blood sugar control, and randomized to either receive the 12 week course of Neulasta (Pegylated granulocyte colony stimulating factor (GCSF)) or a placebo (no medication).

ELIGIBILITY:
Inclusion Criteria:

* Must be > 12 years old and have a confirmed diagnosis of "recent onset T1D" as defined by:
* T1D for < 6 months,
* Stimulated C-peptide ≥ 0.2 pmol/ml
* Presence of at least one diabetes-related autoantibody (e.g., GAD, IA-2, IAA, ICA)
* Normal screening values for CBC
* Willing to comply with intensive diabetes management
* No history of allergy to GCSF
* Females having reproductive potential must be willing to avoid pregnancy and have a negative pregnancy test

Exclusion Criteria:

* Known hypersensitivity to E.Coli-derived proteins, pegfilgrastim, Filgrastim, or any other component of the product
* Chronic use of steroids or other immunosuppressive agents
* Active infection
* Inability to maintain intensive diabetes management
* Pregnancy
* History of malignancy
* Currently participating in another type 1 diabetes treatment study.
* Use of non-insulin pharmaceuticals that affect glycemic control

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve C-peptide Changed Time 0, 12 weeks, 24 weeks, 48 weeks and 96 weeks. | Changed Time 0, 12 weeks, 24 weeks, 48 weeks and 96 weeks.
  The target population distribution of change in the Area Under the Curve in residual beta cell function (C-peptide levels) is the same for treatment and placebo.
Number of participants with adverse events | 96 Weeks

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) levels have the same target distribution for treatment and placebo | 96 weeks
Increase T regulatory cells (Treg) from the bone marrow | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Haller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States